CLINICAL TRIAL: NCT07181187
Title: Phase II Clinical Trial of MH004 Ointment in Patients With Non-segmental Vitiligo
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Minghui Pharmaceutical (Hangzhou) Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MH004-E-201
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- VC Period: MH004 1.0% Ointment QD (Experimental): Participants received MH004 1.0% Ointment once a day (QD) from Day 1 to Week 24 during the Vehicle Control (VC) Period.
  Interventions: Drug: MH004 Ointment
- VC Period: MH004 1.0% Ointment BID (Experimental): Participants received MH004 1.0% Ointment twice daily (BID) from Day 1 to Week 24 during the Vehicle Control (VC) Period.
  Interventions: Drug: MH004 Ointment
- VC Period: Vehicle Ointment QD (Placebo Comparator): Participants received vehicle ointment QD from Day 1 to Week 24 during the VC Period.
  Interventions: Drug: Vehicle Ointment
- VC Period: Vehicle Ointment BID (Placebo Comparator): Participants received vehicle ointment BID from Day 1 to Week 24 during the VC Period.
  Interventions: Drug: Vehicle Ointment
- LTS Period: 1.0% MH004 Ointment QD (Experimental): Participants who completed the Week 24 assessments with no safety concerns could continue into the 28-week Treatment-Extension Period. Participants who applied MH004 1.0% Ointment or Vehicle Ointment QD will apply MH004 1.0% Ointment QD from week 24 to week 52 during the LTS period.
  Interventions: Drug: MH004 Ointment
- LTS Period: 1.0% MH004 Ointment BID (Experimental): Participants who completed the Week 24 assessments with no safety concerns could continue into the 28-week Treatment-Extension Period. Participants who applied MH004 1.0% Ointment or Vehicle Ointment BID will apply MH004 1.0% Ointment BID from week 24 to week 52 during the LTS period.
  Interventions: Drug: MH004 Ointment

INTERVENTIONS:
Drug: MH004 Ointment — MH004 1% ointment applied topically to the affected area as a thin film once or twice daily.
  Arms: LTS Period: 1.0% MH004 Ointment BID; LTS Period: 1.0% MH004 Ointment QD; VC Period: MH004 1.0% Ointment BID; VC Period: MH004 1.0% Ointment QD
Drug: Vehicle Ointment — Matching vehicle ointment applied topically to the affected area as a thin film once or twice daily.
  Arms: VC Period: Vehicle Ointment BID; VC Period: Vehicle Ointment QD

SUMMARY:
This is a multicenter, randomized, double-blind, vehicle-controlled phase II study of MH004 Ointment with a 28-week open-label long-term safety extension period. The study was designed to evaluate the safety, tolerability, pharmacokinetics (PK), and primary efficacy of MH004 Ointment in adolescents and adults with vitiligo.

DETAILED DESCRIPTION:
This phase II trial of MH004 Ointment comprises two periods: a vehicle control period and an open-label long-term safety extension period. Participants will be randomly aligned to the 1.0% MH004 Ointment or Vehicle arms and treated for up to 24 weeks, followed by a 28-week open-label LTS treatment period with 1.0% MH004 Ointment. The primary objective of this trial is to evaluate the efficacy of MH004 Ointment in adolescent and adult participants with vitiligo.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 12 to 65 years (inclusive) of either gender.
2. Clinical diagnosis of non-segmental vitiligo with depigmented area including ≥ 0.5% BSA on the face and total body vitiligo area not exceeding 20% BSA.
3. Fully understand the trial content, voluntarily participate in the trial, and sign the ICF.
4. Must be willing to take appropriate contraceptive measures to avoid pregnancy or fathering a child for the duration of study participation.

   -

Exclusion Criteria:

1. Other dermatoses that may complicate the assessment of vitiligo.
2. Previous depigmentation treatments (eg, monobenzone) for past treatment of vitiligo or other pigmented areas.
3. Use of protocol-defined treatments within the indicated washout period before baseline.
4. Liver or renal damage.
5. Allergic to any component of the investigational drug.
6. Pregnant or lactating subjects. -

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2024-03-26 (Actual); Primary Completion 2025-10-14 (Estimated); Study Completion 2026-05-14 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving Facial Vitiligo Area Scoring Index 50(F-VASI50) at Week 24. | Baseline; Week 24
  An F-VASI50 responder achieved at least 50% improvement from Baseline in F-VASI, measured by the percentage of vitiligo involvement (percentage of body surface area [BSA]) and the degree of depigmentation: 0% (no depigmentation), 10% (only specks of depigmentation), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment), or 100% (no pigment). The percentage of BSA (hand unit) vitiligo involvement was estimated to the nearest 0.1% by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate the percentage of BSA vitiligo involvement. F-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each site on the face and summing the values of all sites (possible range: 0-3; lower scores indicate increased improvement).

SECONDARY OUTCOMES:
Percentage of Participants Achieving a ≥ 75% Improvement from Baseline in the Face Vitiligo Area Scoring Index (F-VASI75) Score at Week 24 | Baseline; Week 24
  An F-VASI75 responder achieved at least 75% improvement from Baseline in F-VASI, measured by the percentage of vitiligo involvement (percentage of body surface area [BSA]) and the degree of depigmentation: 0% (no depigmentation), 10% (only specks of depigmentation), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment), or 100% (no pigment).
Percentage of Participants Achieving a ≥ 50% Improvement from Baseline in the Total Body Vitiligo Area Scoring Index (T-VASI50) Score at Week 24 | Baseline; Week 24
  A T-VASI50 responder achieved at least 50% improvement from Baseline in T-VASI, calculated with contributions from 6 sites. The percentage of vitiligo involvement was estimated in hand units (percentage of BSA estimated to the nearest 0.1%) by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate percent BSA vitiligo involvement. The degree of depigmentation for each site was estimated to the nearest percentage: 0% (no depigmentation present), 10% (only specks of depigmentation present), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment present), 100% (no pigment present). T-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each site and summing the values (range: 0-100; lower scores indicate increased improvement).
Percentage of Participants Achieving a ≥ 75% Improvement from Baseline in the Total Body Vitiligo Area Scoring Index (T-VASI75) Score at Week 24 | Baseline; Week 24
  A T-VASI75 responder achieved at least 75% improvement from Baseline in T-VASI, calculated with contributions from 6 sites
Percentage Change from Baseline in Facial Body Surface Area (F-BSA) at Week 24 | Baseline; Week 24
  F-BSA involvement was the proportion of the facial body surface area with vitiligo. The area "Face" was defined as including the area on the forehead to the original hairline, on the cheek to the jawline vertically to the jawline and laterally from the corner of the mouth to the tragus. The area "Face" did not include surface area of the lips, scalp, ears, or neck, but included the nose and eyelids. Body surface area assessment was performed by the Palmar Method. Body surface area was estimated to the nearest 0.1%. The approximate size of the participant's entire palmar surface (i.e., the palm plus 5 digits) was considered as 1% BSA, and the approximate size of the participant's thumb was considered as 0.1% BSA. Percentage change = ([post-Baseline (BL) value minus BL value]/BL value) X 100.
Percentage Change from Baseline in F-VASI at Week 24 | Baseline; Week 24
  F-VASI was measured by the percentage of vitiligo involvement (percentage of BSA) and the degree of depigmentation: 0% (no depigmentation), 10% (only specks of depigmentation), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment), or 100% (no pigment). The percentage of BSA (hand unit) vitiligo involvement was estimated to the nearest 0.1% by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate the percentage of BSA vitiligo involvement. F-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each site on the face and summing the values of all sites (possible range: 0-3; lower scores indicate increased improvement). Percentage change = ([post-BL value minus BL value]/BL value) X 100.
Percentage Change from Baseline in T-VASI at Week 52 | Baseline; Week 52
  T-VASI was calculated with contributions from 6 sites. The percentage of vitiligo involvement was estimated in hand units (percentage of BSA estimated to nearest 0.1%) by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate percent BSA vitiligo involvement. The degree of depigmentation for each site was estimated to the nearest percentage: 0% (no depigmentation present), 10% (only specks of depigmentation present), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment present), 100% (no pigment present). T-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each site and summing the values (range: 0-100; lower scores indicate increased improvement). Percentage change = ([post-BL value minus BL value]/BL value) X 100.
Proportion of participants achieving Facial Vitiligo Area Scoring Index 50(F-VASI50) at Week 52. | Baseline; Week 52
  An F-VASI50 responder achieved at least 50% improvement from Baseline in F-VASI, measured by the percentage of vitiligo involvement (percentage of body surface area [BSA]) and the degree of depigmentation: 0% (no depigmentation), 10% (only specks of depigmentation), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment), or 100% (no pigment).
Percentage of Participants Achieving a ≥ 50% Improvement from Baseline in the Total Body Vitiligo Area Scoring Index (T-VASI50) Score at Week 52 | Baseline; Week 52
  A T-VASI50 responder achieved at least 50% improvement from Baseline in T-VASI, calculated with contributions from 6 sites.
Percentage Change From Baseline in T-BSA at Week 52 | Baseline; Week 52
  T-BSA involvement was the proportion of the body surface area with vitiligo. Body surface area assessment was performed by the Palmar Method. Body surface area was estimated to the nearest 0.1%. The approximate size of the participant's entire palmar surface (i.e., the palm plus 5 digits) was considered as 1% BSA, and the approximate size of the participant's thumb was considered as 0.1% BSA. Percentage change = ([post-BL value minus BL value]/BL value) X 100.
Number of Participants With Treatment-emergent Adverse Events (TEAEs) | From the time of Informed Consent Form signing until at least 30 days after the last application of study drug (up to Week 52)
  An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug-related. An AE could have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study treatment. A TEAE was defined as any AE reported for the first time or the worsening of a pre-existing event after the first application of study drug.

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou Third People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No